CLINICAL TRIAL: NCT05567315
Title: Interest of Hypnosis in Virtual Reality on Nociception During Oocyte Retrieval in a Medically Assisted Reproduction Procedure: a Randomised Controlled Study
Brief Title: Interest of Hypnosis in Virtual Reality on Nociception During Oocyte Retrieval in a Medically Assisted Reproduction Procedure
Acronym: HypnoPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Mutualiste la Sagesse (Other)
Responsible Party: Principal Investigator, Vincent Denoual, Anesthesiologist, Clinique Mutualiste la Sagesse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-A02136-35
Record Dates: First submitted 2022-02-24; First posted 2022-10-05 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Oocyte Retrieval
MeSH Terms: interventions — Anesthesia, Local; Hypnosis

STUDY DESIGN:
Intervention Model Description: Single-centre, comparative, randomised, parallel group study
Who Masked: Outcomes Assessor
Masking Description: The person collecting the endpoints will be blinded to the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oocyte puncture with local anaesthesia alone (Active Comparator)
  Interventions: Drug: local anaesthetic injection
- Oocyte puncture with local anaesthesia and additional virtual reality hypnosis (Experimental)
  Interventions: Drug: local anaesthetic injection; Device: hypnosis with Virtual reality mask

INTERVENTIONS:
Drug: local anaesthetic injection — Infiltration of 40 to 80 ml of a non-adrenalized 0.5% lidocaine solution into the vaginal wall at the level of the vaginal pouches, under ultrasound guidance. (within the limit of the toxic doses, i.e. 5mg/kg)
Device: hypnosis with Virtual reality mask — A 20-minute virtual reality hypnosis session is performed from the time the patient is placed on the surgical table until the end of the oocyte poncture
  Arms: Oocyte puncture with local anaesthesia and additional virtual reality hypnosis

SUMMARY:
Study on the effect of the virtual hypnosis mask in addition to local anaesthesia on anxiety and perioperative pain during oocyte puncture

ELIGIBILITY:
Inclusion Criteria:

* Patient having an oocyte puncture as part of a medically assisted procreation procedure
* Surgical procedure planned in the operating theatre under local anaesthesia at the Clinique Mutualiste La Sagesse
* Patient capable of receiving and understanding information about the study and giving written informed consent.
* Affiliated to a social security system

Exclusion Criteria:

* Patient's refusal to participate in a study
* Patient having an oocyte retrieval as part of an oocyte donation
* Unbalanced epilepsy.
* Hearing and/or visual impairments that contraindicate the use of the virtual reality headset.
* Patient with a poor understanding of the French language.
* Medical indication to carry out the oocyte puncture under general anaesthesia
* Drug allergy or hypersensitivity to PARACETAMOL - IBUPROFEN or NEFOPAM prescribed during the pre-medication.
* Patient under legal protection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 182 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Analgesia Nociception Index (ANI) measurement | during oocyte puncture procedure
  The level of pain perceived by the patient during the performance of a painful care procedure will be measured by the ANI index which reflects heart rate variability

SECONDARY OUTCOMES:
Anxiety with beck anxiety inventory | 1 hour before intervention and immediately after the intervention
  Measurement of anxiety by the Beck Anxiety Inventory, on admission to hospital and on return to the ward, 1 hour after the oocyte puncture
Simulator Sickness Questionnaire (SSQ) | Immediately after the intervention
  Assessment of tolerance of virtual reality with SSQ ; SSQ is a scale of cyber sickness from 0 to 48, a higher score mean a worse outcome.
Analog visual scale (AVS) | Immediately after the intervention
  Pain evaluation with Analog visual scale by the patient himself from 0 to 10, a higher score mean a worse outcome.
Post intervention analgesic therapy | Immediately after the intervention
  Identify the need for postoperative analgesic treatment in the two groups
Total duration of the procedure of oocyte ponction (min) | From the first ponction of local anesthesia to the end of the retrieval of the last oocyte
  Total duration of the procedure (min), from the beginning of local anesthesia to the end of the oocyte retrieval
Conversion rate from local anaesthesia to unplanned general anaesthesia | Immediately after the intervention
  Conversion rate in percent
Gynecologist's numerical satisfaction scale | Immediately after the intervention
  Measure by a numerical scale out of 10, a higher score mean a better outcome.
Patient's numerical satisfaction scale | Immediately after the intervention
  Measure by a numerical scale out of 10, a higher score mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique mutualiste La Sagesse, Rennes, Brittany Region, France